CLINICAL TRIAL: NCT05576922
Title: Xenogeneic Collagen Matrix Loaded With rhPDGF-BB vs Autogenous Connective Tissue Graft for the Treatment of Peri-implant Soft Tissue Dehiscences: A Randomized, Controlled, Clinical, Trial
Brief Title: Collagen Matrix + rhPDGF-BB vs Connective Tissue Graft for the Treatment of Peri-implant Soft Tissue Dehiscences
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Lorenzo Tavelli, Principal Investigator, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Delta IMPL REC (IRB22-0637)
Record Dates: First submitted 2022-10-03; First posted 2022-10-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Implant Complication
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Intervention Model Description: Parallel-arm
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Connective tissue graft (Active Comparator): Autogenous connective tissue graft harvested from the palate as a free gingival graft and then de-epithelialized
  Interventions: Other: Prosthetic-surgical approach + autogenous graft
- Collagen matrix + rhPDGF-BB (Experimental): Xenogeneic cross-linked collagen matrix + recombinant human platelet-derived growth factor-BB
  Interventions: Other: Prosthetic-surgical approach + graft substitute

INTERVENTIONS:
Other: Prosthetic-surgical approach + autogenous graft — Coronally advanced flap with an autogenous graft (CTG)
  Arms: Connective tissue graft
Other: Prosthetic-surgical approach + graft substitute — Coronally advanced flap with a graft substitute (collagen matrix and rhPDGF-BB)
  Arms: Collagen matrix + rhPDGF-BB

SUMMARY:
The study aims at comparing two different approaches for the treatment of implant esthetic complications (peri-implant soft tissue dehiscences): autogenous connective tissue graft vs collagen matrix + recombinant human platelet derived growth factor-BB

DETAILED DESCRIPTION:
The present randomized clinical trial aims at investigating two approaches (autogenous connective tissue graft vs collagen matrix + recombinant human platelet derived growth factor-BB) when performed in combination with the prosthetic-surgical approach for the treatment of peri-implant soft tissue dehiscences. Clinical, volumetric, ultrasonographic and patient-reported outcomes will be evaluated at different time points up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Periodontally and systemically healthy,
* Full-mouth plaque score and full-mouth bleeding score ≤ 20% (measured at four sites per tooth), iv) Presence of single dental implant in the anterior area (from the first right premolar to the first left premolar) showing a PSTD, with the subjects searching for treatment of this condition,
* Peri-implant papillae not flat (PSTD subclass a or b) (Zucchelli et al., 2019), vi) Implants diagnosed as healthy (Berglundh et al., 2018),
* Ability to perform good oral hygiene

Exclusion Criteria:

* Contraindications for surgery,
* Systemic condition (e.g. diabetes mellitus, HIV, cancer, etc) that could compromise wound healing,
* Patients pregnant or attempting to get pregnant (self-reported),
* Untreated periodontitis,
* Untreated peri-implant mucositis or peri-implantitis (Berglundh et al., 2018),
* Smoking, defined as self-reported daily habit. Occasional smokers won't be excluded,
* History of soft tissue grafting at the implant site showing PSTD within the last 6 months.

Indications for surgical intervention will be established based on patient's esthetic demands and peri-implant soft tissue phenotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Soft tissue dehiscence reduction | 6 and 12 months
  Reduction of the depth of the Soft tissue dehiscence (vertical measurement of the complication, in relation to the level of the cemento-enamel junction of the contralateral homologous tooth) compared to baseline (expressed in millimeters)

SECONDARY OUTCOMES:
Complete peri-implant soft tissue dehiscence (PSTD) coverage | 6 and 12 months
  Percentage of cases with complete resolution of the implant esthetic complication (expressed as a percentage)
mean peri-implant soft tissue dehiscence (PSTD) coverage | 6 and 12 months
  Percentage of coverage of the soft tissue dehiscence compared to baseline, measured with a formula considering final PSTD depth and initial PSTD depth (expressed as a percentage)
Mucosal thickness changes | 3, 6 and 12 months
  Changes within the mucosal thickness measured with ultrasonography (expressed in mm)
3D Volumetric changes | 3, 6 and 12 months
  Changes within the buccal contour measured by superimposing digital impressions obtained with optical scanning (expressed in mm^3)
Post-operative pain | 14 days after the surgery
  Patient-reported pain after the surgical procedure (expressed with a 0-10 visual analogue scale [VAS])
Professional esthetic assessment | 12 months
  Esthetic outcomes of the treatment assessed by a calibrated operator using the Implant soft tissue Dehiscence coverage Esthetic Score (IDES) (expressed using points, based on the IDES classification system from Zucchelli et al. 2021)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Tavelli, DDS, MS, Principal Investigator — Harvard School of Dental Medicine, Boston, USA
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No